CLINICAL TRIAL: NCT03169192
Title: Molecular Genetic Study of Suspected Cases of Osteogenesis Imperfecta Attending Assiut University Children Hospital
Brief Title: Diagnosis of Osteogenesis Imperfecta in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mohamed aboubakr mohamed, principal investigator, Assiut University
Other Study IDs: OI
Record Dates: First submitted 2017-05-25; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Bone Disease, Metabolic
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Zoledronic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — we collect blood samples of patients to detect COLLAGEN I AI gene and COLLAGEN 1 A2 gene
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Repeated fractures group: detection of gene mutations of osteogenesis imperfecta in single group of patients with repeated fractures then start treatment with zoledronic acid in doses children less than 5 years ( 0.025 milligram for each kilogram every 3 months for 18 months duration) children more than 5 years ( 0.05 milligram for each kilogram every 6 months for 18 months duration)
  Interventions: Drug: Zoledronic Acid

INTERVENTIONS:
Drug: Zoledronic Acid — intravenous injections once every 3 months

SUMMARY:
The study will be conducted at Assiut university children hospital and it will include patients with history of repeated fractures due to mild or irrelevant trauma.

Diagnosis will be established by biochemical tests, bone survey to exclude secondary causes followed by Dual Energy absorbiometry scan to detect bone density of selected cases then confirm our diagnosis by detection of gene mutations of Osteogenesis imperfecta during one and half year duration with starting zoledronic acid therapy during this duration.

DETAILED DESCRIPTION:
Osteogenesis imperfecta is a genetic disorder of the connective tissue matrix caused by abnormal collagen microﬁbril assembly, .Several clinical subtypes of Osteogenesis imperfecta have been described based on the clinical, biochemical, and molecular nature of the disorder . New research is emphasizing the structural interaction within the microﬁbril and identifying regions within the collagen, which play greater or lesser roles in the structural properties of the triple helix, .In taking this information into account, clinical phenotypes resulting from certain mutations can be predicted because of this pathogenetic correlation.

The clinical manifestations vary considerably, ranging from a severe perinatal lethal form to a mild disorder which only becomes evident in adulthood, manifesting as premature osteoporosis, .Most commonly, however, Osteogenesis imperfecta presents in childhood with multiple fractures and related complications, .The precise incidence of Osteogenesis imperfecta is unknown and reports vary from approximately 1/100,000 to 1/25,000 dependent on the criterion used to deﬁne Osteogenesis imperfecta.

Severe forms and milder disease occur with approximately similar incidence. Severe and mild forms share the cardinal feature of bone fragility, which is characterized by bone fractures often after little or no trauma, .Several ﬁndings in Osteogenesis imperfecta are common to other disorders of connective tissues; hyper-mobile joints and a blue sclera are among these features frequently described, The incorporation of abnormal type 1 collagen in teeth results in brittle opalescent teeth, the hallmark of Dentinogenesis Imperfecta, often seen in Osteogenesis imperfecta, .Progressive conductive hearing loss in early adulthood is the result of damage to the ossicles in the middle ear; over time, hearing loss typically progresses and combined conductive and sensorineural hearing loss may be seen in adults, similar to that of otosclerosis. Short stature and bone deformity are common features of the disorder The mainstay of treatment is orthopedic management along with physiotherapy, Bisphosphonates are being evaluated for efﬁcacy and clinical trials have shown improvement at least in bone mineral density

Disorders associated with fragility fractures in children:

A) Primary conditions

1. Genetic disorders :- Osteogenesis imperfecta - Ehlers-Danlos syndrome - Marfan syndrome Homocystinuria - Osteoporosis - Hypophosphatasia Polyostotic fibrous dysplasia - Rickets (genetic forms)
2. Idiopathic juvenile osteoporosis B) Secondary conditions

1- Chronic inflammatory conditions Systemic lupus erythematosus - Inflammatory bowel disease - Nephrotic syndrome 2- Reduced mobility Cerebral palsy - Duchenne muscular dystrophy - Posttraumatic 3- Infiltrative Leukemia - Thalassemia

4- Endocrine Hypogonadism - Growth hormone deficiency - Cushing syndrome Hyperthyroidism - Diabetes mellitus 5- Nutritional/malabsorptive Vitamin D deficiency - Celiac disease - Biliary atresia Cystic fibrosis - Anorexia nervosa 6- Renal Chronic kidney disease - Secondary hyperparathyroidism 7- Iatrogenic Glucocorticoids - Anticonvulsants - Methotrexate - Radiation therapy

ELIGIBILITY:
Inclusion Criteria:

1. Positive family history of fractures or stillbirths.
2. Results of biochemical tests correlate with osteogenesis imperfecta.
3. Low bone density.

Exclusion Criteria:

1. Presence of secondary causes of fractures.
2. Abnormalities of biochemical tests or hormonal profile.
3. Negative family history.
4. Fractures in same site each time.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Any Infants or children from age of 1 month up to age of 18 years presented with History of repeated fractures (more than one)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of children diagnosed as osteogenesis imperfecta | 1 month
  diagnosis based on molecular genetic study

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Folkestad L, Hald JD, Hansen S, Gram J, Langdahl B, Abrahamsen B, Brixen K. Bone geometry, density, and microarchitecture in the distal radius and tibia in adults with osteogenesis imperfecta type I assessed by high-resolution pQCT. J Bone Miner Res. 2012 Jun;27(6):1405-12. doi: 10.1002/jbmr.1592. PMID 22407910
- [Result] Cheung MS, Glorieux FH. Osteogenesis Imperfecta: update on presentation and management. Rev Endocr Metab Disord. 2008 Jun;9(2):153-60. doi: 10.1007/s11154-008-9074-4. Epub 2008 Apr 11. PMID 18404382
- [Result] Bachrach LK, Gordon CM; SECTION ON ENDOCRINOLOGY. Bone Densitometry in Children and Adolescents. Pediatrics. 2016 Oct;138(4):e20162398. doi: 10.1542/peds.2016-2398. PMID 27669735
- [Result] Phillipi CA, Remmington T, Steiner RD. Bisphosphonate therapy for osteogenesis imperfecta. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD005088. doi: 10.1002/14651858.CD005088.pub2. PMID 18843680